CLINICAL TRIAL: NCT07105241
Title: Virtual Reality in Electrophysiological Procedures and Device Implantation: the VR inEP Trial
Acronym: VR inEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL-010331
Record Dates: First submitted 2025-07-10; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Arrhythmia; Cardiac Implantable Electronic Device; Ablation of Arrhythmias; Electrophysiologic Study; Pacemaker; ICD
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR therapy (Experimental)
  Interventions: Other: VR therapy; Other: 360 degree education videos
- Control group (No Intervention): The control group is treated according to the local protocol, which may encompass preprocedural administration of benzodiazepines or analgesics depending on the procedure type and indication, nurses' assessment, patient preference, comorbidities, and medication use. These medications will be administered after randomization and baseline assessment of anxiety and pain. If required during the procedure, additional analgesics may be administered (usually fentanyl).

INTERVENTIONS:
Other: VR therapy — Patients in the VR intervention group receive a VR 'relax and distract' intervention in addition to standard care. This type of VR utilizes video's, relaxation exercises and cognitive games to immerse patients in a novel, calming and distracting environment, enhancing the patient's ability to manage anxiety, stress and pain. The VR set is introduced to the patient in the cardiology day care unit prior to the procedure allowing for familiarization with the device. After moving the patient to the catheterization laboratory, the VR set is re-offered to the patient and the VR intervention is started. The intervention ends with the conclusion of the procedure, or when the patient indicates that they would like to discontinue the therapy earlier.
  Other Names: VR relax and distract; VR relax & distract; Virtual reality
  Arms: VR therapy
Other: 360 degree education videos — Prior to the procedure, patients in the VR intervention group are additionally offered an educational video consisting of a virtual tour of the EP laboratory with a visual explanation of the upcoming procedure. These videos will be recorded as 360ͦ videos to support an optimal immersive experience when viewed on the VR set. In this way, the videos will serve simultaneously as additional educational measures for the procedure, as well as a way to familiarize patients with the VR set. Use of the educational videos is not obligatory, but is offered optionally according to patients' preference.
  Arms: VR therapy

SUMMARY:
Each year about 37,000 patients undergo a catheter ablation to treat cardiac arrhythmias or have a cardiac device such as a pacemaker or implantable cardioverter defibrillator implanted in the Netherlands. Although the procedures positively impact health related outcomes on the long term, they are often accompanied by periprocedural pain and anxiety on a shorter term. These negative effects can be prevented or treated by pharmacological interventions (e.g. analgesics or benzodiazepines), but side effects of these drugs may compromise patient safety and extend hospital admissions. Distraction using Virtual Reality (VR) may be an attractive non-pharmacological alternative.

It is the aim of the Virtual Reality in Electrophysiological Procedures and device implantation (VR inEP) trial to study the feasibility and efficacy of VR to decrease experienced pain and anxiety in patients undergoing invasive procedures for arrhythmias and conduction disorders. The study also serves as a stepping stone towards structural implementation of VR into clinical care, by familiarizing care personnel of the cardiac catheterization rooms with the use of VR, its indications and logistics, and identifying potential barriers for structural implementation of VR.

VR inEP is a single-center, open label, randomized controlled trial performed in the catheterization rooms in the Radboudumc. Adult patients undergoing an electrophysiological procedure (e.g., catheter ablation or electrophysiological study) or cardiac device implantation (e.g., pacemaker or implantable cardioverter defibrillator) performed under local anesthesia are eligible for inclusion. Patients consenting to participate are randomized in a 1:1 ratio to the VR intervention or control group, stratified for the indication for the procedure (50% electrophysiological procedures, 50% cardiac device implantations). Patients and their treatment teams are unblinded for the treatment allocation. The primary outcomes are pain perception and anxiety during the procedure as a whole, quantified using the visual analog scale (VAS) for pain and the numeric ranking scale (NRS) for anxiety, 30 minutes after the procedure ends.

DETAILED DESCRIPTION:
Rationale: Each year approximately 37,000 patients undergo a catheter ablation or cardiac device implantation in The Netherlands. Although the procedures positively impact health related outcomes, they are often accompanied by periprocedural pain and anxiety. These negative effects can be prevented or treated by pharmacological interventions (e.g. analgesics or benzodiazepines), but side effects of these drugs may compromise patient safety and extend hospital admissions. Distraction using Virtual Reality (VR) may be an attractive non-pharmacological alternative.

Objective: it is the aim of the Virtual Reality in Electrophysiological Procedures and device implantation (VR inEP) trial to study the feasibility and efficacy of VR to decrease experienced pain and anxiety in patients undergoing invasive procedures for arrhythmias and conduction disorders. The study also serves as a stepping stone towards structural implementation of VR into clinical care, by familiarizing care personnel of the cardiac catheterization rooms with the use of VR, its indications and logistics, and identifying potential barriers for structural implementation of VR.

Study design: VR inEP is a single-center, open label, randomized controlled trial performed in the catheterization rooms in the Radboudumc.

Study population: Adult patients undergoing an electrophysiological procedure (e.g., catheter ablation or electrophysiological study) or cardiac device implantation (e.g., pacemaker or implantable cardioverter defibrillator) performed under local anesthesia are eligible for inclusion.

Intervention: Patients consenting to participate are randomized in a 1:1 ratio to the VR intervention or control group, stratified for the indication for the procedure (50% electrophysiological procedures, 50% cardiac device implantations). Patients and their treatment teams are unblinded for the treatment allocation.

Main study parameters: The primary outcomes are pain perception and anxiety during the procedure as a whole, quantified using the visual analogue scale (VAS) for pain and the numeric ranking scale (NRS) for anxiety, 30 minutes after the procedure ends.

ELIGIBILITY:
Inclusion Criteria:

* ≥16 years of age
* Planned to undergo an invasive electrophysiological procedure (e.g., catheter ablation or electrophysiological study) or cardiac device implantation (e.g., pacemaker or implantable cardioverter defibrillator).
* The procedure must be performed under local anesthesia.

Exclusion Criteria:

* Patients undergoing procedures using (conscious) sedation
* Patients who do not speak or understand Dutch
* History of dementia
* Severe visual impairment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain perception | 0.5-6 hours
  Pain perception during the procedure as a whole, quantified using the visual analogue scale (VAS, 0-10 points) 30 minutes after the procedure ends.
Anxiety | 0.5-6 hours
  The second primary outcome is anxiety during the procedure as a whole, quantified using the numeric ranking scale (NRS, 0-10 points) 30 minutes after the procedure ends.

SECONDARY OUTCOMES:
Use of analgesics | 0.5-6 hours
Self-reported acceptable pain | 0.5-6 hours
  Self-reported answer, provided in custom made questionnaire (yes/no)
Worst pain | 0.5-6 hours
  Measured on the Visual Analogue Scale
Time experience | 0.5-6 hours
  Self-reported answer by patients, provided in custom made questionnaire (expected number of hours/minutes duration of the procedure)
Heart rate variability | 0.5-6 hours
Procedural duration | 0.5-6 hours
Duration of hospital admission after finalization of the procedure | 0-7 days
Time of VR use as a percentage of total procedural duration | 0.5-6 hours
Patient satisfaction with the VR therapy and the optional educational video | 0.5-10 hours
  Score from 0-10, where 10 is the highest value/satisfaction
Procedural satisfaction of health care professionals with VR | 0.5-10 hours
  Satisfaction score from 0-10, where 10 is the highest value/satisfaction
Number of patients with complications | 0.5-6 hours

IPD SHARING:
Plan to Share IPD: Undecided